CLINICAL TRIAL: NCT01250080
Title: Effect of Gutamine Administration in the Innate Immune System Response in ICU Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Espen (Other); This research prize was funded by Nestle Nutrition Institute and by Fresenius Kabi. (Unknown)
Responsible Party: Jon Pérez Bárcena, Hospital Universitari Son Dureta
Allocation: Randomized | Masking: Single
Other Study IDs: IB709/06
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-09

CONDITIONS: Moderate to Severe Trauma, as Defined by an; Injury Severity Score (ISS) > 12 Points Were Included in the Study.
MeSH Terms: interventions — Parenteral Nutrition, Total; Glutamine

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Glutamine (Experimental)
  Interventions: Dietary Supplement: Total Parenteral Nutrition with Glutamine
- Control (Sham Comparator)
  Interventions: Other: Total Parenteral Nutrition without glutamine

INTERVENTIONS:
Dietary Supplement: Total Parenteral Nutrition with Glutamine — daily glutamine supplement of 0.35 g/kg weight as N2-L-Alanyl-L-Glutamine (0.5 g/kg/d - Dipeptiven Fresenius Kabi España) during five days.
  Arms: Glutamine
Other: Total Parenteral Nutrition without glutamine — The control group received a supplemental volume of the basic TPN solution to achieve an isocaloric an isonitrogenated formula with the study group.
  Arms: Control

SUMMARY:
Glutamine is the most abundant nonessential amino acid in the human body. Besides its role as a constituent of proteins and its importance in amino acid transamination, glutamine may modulate immune cells.

The innate immune system is the first line of host defence against pathogens and in most cases sufficient to eliminate invading microbes. Mammalian Toll-like receptors (TLR) comprise a family of germ line-encoded trans-membrane receptors which activation leads to the induction of inflammatory responses, phagocytosis but also to the development of antigen specific adapative immunity.

It has been postulated though not formally proven yet that glutamine beneficial effect could be due to a positive effect on the innate immune system. Given the importance of TLRs and TLRs-dependent signalling in host defence against infections we hypothesized that glutamine may increase the expression and/or functionality of TLRs which in turn may have beneficial effects to clear infections.

DETAILED DESCRIPTION:
Objective: To evaluate whether glutamine supplementation alters the expression and functionality of TLR2 and TLR4 in circulating monocytes of trauma patients admitted to the ICU. Specifically the next variables were measured:

* Expression of TLR2 and TLR4 in peripheral blood monocytes was determined by flow cytometry
* To study the functionality of TLR2 and TLR4, monocytes were stimulated with TLR specific agonists and cytokines were measured in cell culture supernatants. We determined the concentration of IL-1β, IL-6, TNFα and IL-10 in cell culture supernatants using a bead array ELISA.
* To determine the phagocytic capability of monocytes, live Escherichia coli expressing green fluorescent protein was added to 100 μL of whole blood collected in K2-anticoagulation medium tubes. Bacteria were added at a ratio of 100 bacteria per monocyte. The analyses were carried out in an Epics XL flow cytometer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years (inclusive).
* Moderate to severe trauma, as defined by an Injury Severity Score (ISS) > 12 points were included in the study
* Traumatic patients who required total parenteral nutrition

Exclusion Criteria:

* Patients who were under 17 and over 76 years of age,
* Patients whose life expectancy was less than 5 days
* Patientes allergic to glutamine.
* Patients with any basic pathology included any serious immune system condition (diabetes, HIV, lupus, etc.) or who, in their long-term treatment prior to admission to ICU, received corticoids or any other immunosuppressant medication.
* Pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
-Expression of TLR2 and TLR4 in peripheral blood monocytes was determined by flow cytometry

SECONDARY OUTCOMES:
-To study the functionality of TLR2 and TLR4, monocytes were stimulated with TLR specific agonists and cytokines were measured in cell culture supernatants.
- To determine the phagocytic capability of monocytes, live Escherichia coli expressing green fluorescent protein was added to 100 μL of whole blood collected in K2-anticoagulation medium tubes.

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit. Hospital Universitario Son Dureta, Palma Mallorca, Balearic Islands, Spain

REFERENCES:
- [Derived] Perez-Barcena J, Crespi C, Regueiro V, Marse P, Raurich JM, Ibanez J, Garcia de Lorenzo-Mateos A, Bengoechea JA. Lack of effect of glutamine administration to boost the innate immune system response in trauma patients in the intensive care unit. Crit Care. 2010;14(6):R233. doi: 10.1186/cc9388. Epub 2010 Dec 24. PMID 21184675